CLINICAL TRIAL: NCT06353087
Title: The Real-world Treatment Patterns and Clinical Outcomes in Moderate-to-severe Atopic Dermatitis (AD) Patients Receiving Abrocitinib
Brief Title: Abrocitinib Taiwan Treatment Pattern and Real World Study in ATopiC Dermatitis (ATTRACT Registry)
Acronym: ATTRACT
Status: Recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B7451114; NCT06353087 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-03-21; First posted 2024-04-08 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Dermatitis, Atopic; Dermatitis; Eczema; Skin Diseases; Immune System Diseases; Janus Kinase Inhibitors
Keywords: Atopic Dermatitis; Abrocitinib; JAK inhibitors; Real world; Registry; Taiwan
MeSH Terms: conditions — Dermatitis, Atopic; Dermatitis; Eczema; Skin Diseases; Immune System Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is to describe the real-world treatment patterns and clinical outcomes in moderate-to-severe AD patients receiving abrocitinib over a 12-month observation period, and to describe patient demographic and baseline characteristics.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Patients aged ≥12 years
2. Patients with confirmed diagnosis of moderate-to-severe AD as assessed by the physician
3. Patients for whom the physician's decision has been made to newly prescribe abrocitinib in usual clinical practice conditions
4. Evidence of a personally signed and dated informed consent/assent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study

Exclusion Criteria:

Patients meeting any of the following criteria will not be included in the study:

1. Any prior use of abrocitinib
2. Simultaneous participation in a study that includes administration of any investigational drug or procedure

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric AD patients ≥12 years with moderate-to-severe atopic dermatitis receiving abrocitinib.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving >= 75% Improvement From Baseline in Eczema Area and Severity Index (EASI-75) Response at Week 2, 12, 52 | Week 2, 12, 52
  EASI quantifies severity of AD based on severity of lesion clinical signs and percentage (%) of body surface area (BSA) affected. Severity of clinical signs of AD lesions (erythema, induration/papulation, excoriation and lichenification) were scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin)] and lower limbs [including buttocks]) on a 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based on % BSA with AD in body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score ranged from 0.0 to 72.0, with higher scores indicating greater severity of AD.
Percentage of Participants Achieving >= 90% Improvement From Baseline in Eczema Area and Severity Index (EASI-90) Response at Week 2, 12, 52 | Week 2, 12, 52
  EASI quantifies severity of AD based on severity of lesion clinical signs and percentage (%) of body surface area (BSA) affected. Severity of clinical signs of AD lesions (erythema, induration/papulation, excoriation and lichenification) were scored separately for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin)] and lower limbs [including buttocks]) on a 4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based on % BSA with AD in body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score ranged from 0.0 to 72.0, with higher scores indicating greater severity of AD.
Percentage of Participants Achieving Investigator's Global Assessment (IGA) Response of Clear (0) or Almost Clear (1) and Greater Than or Equal to 2 Points Improvement From Baseline at Week 2, 12, 52 | Week 2, 12, 52
  IGA assesses severity of AD on a 5 point scale (0 to 4, higher scores indicate more severity). Scores: 0= clear, no inflammatory signs of AD; 1= almost clear, AD not fully cleared- light pink residual lesions (except post-inflammatory hyperpigmentation), just perceptible erythema, papulation/induration lichenification, excoriation, and no oozing/crusting; 2= mild AD with light red lesions, slight but definite erythema, papulation/induration, lichenification, excoriation and no oozing/crusting; 3= moderate AD with red lesions, moderate erythema, papulation/induration, lichenification, excoriation and slight oozing/crusting; 4= severe AD with deep dark red lesions, severe erythema, papulation/induration, lichenification, excoriation and moderate to severe oozing/crusting. Assessment excluded sole, palms and scalp.

SECONDARY OUTCOMES:
Duration of Abrocitinib Treatment: All Participants | During post-index period (12 months duration post index date)
  Duration of treatment with abrocitinib was the time from date of start of abrocitinib treatment to date of end of abrocitinib treatment or of latest follow-up if not suspended.
Demographic and baseline characteristics | During pre-index period
Percent Change From Baseline in Eczema Area and Severity Index (EASI) Total Score at Week 2, 4, 12, 16, 24, and 52 | Baseline, Week 2, 4, 12, 16, 24, and 52
  EASI evaluates severity of participant's AD (excluded scalp, palms, soles) based on severity of AD clinical signs and % of body surface area (BSA) affected. Severity of clinical signs of AD (erythema, induration/papulation, excoriation and lichenification) scored separately for each of 4 body regions(head and neck, upper limbs, trunk [including axillae and groin] and lower limbs [including buttocks]) on4-point scale: 0= absent; 1= mild; 2= moderate; 3= severe. EASI area score was based upon % BSA with AD in each 4 body region: 0 (0%), 1 (>0 to <10%), 2 (10 to <30%), 3 (30 to <50%), 4 (50 to <70%), 5 (70 to <90%) and 6 (90 to 100%). Total EASI score =0.1*Ah*(Eh+Ih+Exh+Lh) + 0.2*Au*(Eu+Iu+ExU+Lu) + 0.3*At*(Et+It+Ext+Lt) + 0.4*Al*(El+Il+Exl+Ll); A = EASI area score; E = erythema; I = induration/papulation; Ex = excoriation; L = lichenification; h = head and neck; u = upper limbs; t = trunk; l = lower limbs. Total EASI score ranged from 0.0 to 72.0, higher scores = greater severity of AD.
Change From Baseline in Investigator's Global Assessment (IGA) at Weeks 2, 4, 12, 16, 24, and 52 | Baseline, Week 2, 4, 12, 16, 24, and 52
  IGA assesses severity of participant's AD on a 5 point scale. 0= clear, no inflammatory signs of AD; 1= almost clear, AD not fully cleared- light pink residual lesions (except post-inflammatory hyperpigmentation), just perceptible erythema, papulation/induration lichenification, excoriation, and no oozing/crusting; 2= mild AD with light red lesions, slight but definite erythema, papulation/induration, lichenification, excoriation and no oozing/crusting; 3= moderate AD with red lesions, moderate erythema, papulation/induration, lichenification, excoriation and slight oozing/crusting and 4= severe AD with deep dark red lesions, severe erythema, papulation/induration, lichenification, excoriation and moderate to severe oozing/crusting. Higher scores indicating more severity of AD. Assessment excluded soles, palms and scalp.
Change From Baseline in Percentage Body Surface Area at Week 2, 4, 12, 16, 24, and 52 | Baseline, Week 2, 4, 12, 16, 24, and 52
  4 body regions were evaluated: head and neck, upper limbs, trunk (including axillae and groin) and lower limbs (including buttocks). Scalp, palms and soles were excluded. BSA was calculated using handprint method. Number of handprints (size of participant's hand with fingers in a closed position) fitting in the affected area of a body region was estimated. Maximum number of handprints were 10 for head and neck, 20 for upper limbs, 30 for trunk and 40 for lower limbs. Surface area of body region equivalent to 1 handprint: 1 handprint was equal to 10% for head and neck, 5% for upper limbs, 3.33% for trunk and 2.5% for lower limbs. Percent BSA for a body region was calculated as = total number of handprints in a body region * % surface area equivalent to 1 handprint. Overall % BSA for an individual: arithmetic mean of % BSA of all 4 body regions, ranges from 0 to 100%, with higher values representing greater severity of AD.
Change From Baseline in Patient-Oriented Eczema Measure (POEM) at Week 2, 4, 12, and 52 | Baseline, Week 2, 4, 12, and 52
  POEM is a 7-item participant reported outcome (PRO) measure used to assess the impact of AD (dryness, itching, flaking, cracking, sleep loss, bleeding and weeping) over the past week. Each item is scored as "no days (0)", "1-2 days (1)", "3-4 days (2)", "5-6 days (3)" and "every day (4)". The score ranges from 0 to 28, where higher score indicated greater severity.
Change from baseline of Atopic Dermatitis Control Tool (ADCT) score at Week 2, 4, 12, and 52 | Baseline, Week 2, 4, 12, and 52
  The Atopic Dermatitis Control Tool (ADCT) is a brief patient self-administered instrument designed and validated to assess patient-perceived AD control; AD symptoms and impacts are evaluated over the past week, including overall severity of symptoms, days with intense episodes of itching, intensity of bother, problem with sleep, impact on daily activities, and impact on mood or emotions
Change From Baseline in Dermatology Life Quality Index (DLQI) Total Score to Week 2, 4, 12, and 52 | Baseline, Week 2, 4, 12, and 52
  The DLQI was a 10-item questionnaire that measures the impact of skin disease on participant's quality of life. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicate more impact on quality of life. The DLQI total score ranges from 0 (not at all) to 30 (very much): 0-1 = no effect at all on the participant's life; 2-6 = small effect on the participant's life; 7-12 = moderate effect on the participant's life; 13-18 = very large effect on the participant's life; 19-30 = extremely large effect on the participant's life. Higher scores indicate more impact on quality of life of participants.
Change From Baseline in Patient Global Assessment (PtGA) | Baseline, Week 2, 4, 12, 16, 24, and 52
  The PtGA asked the participant to evaluate the overall cutaneous disease at that point in time on a single-item, 5-point scale. The same category labels used in the IGA were used for the PtGA, ie, "severe (4)", "moderate (3)", "mild (2)","almost clear (1)", and "clear (0)". The PtGA was completed as per schedule of activities.
Percentage Change From Baseline in Peak Pruritus Numerical Rating Scale (PP-NRS) From Baseline at Weeks 2, 4, 12, 16, 24, and 52 | Baseline, Week 2, 4, 12, 16, 24, and 52
  The severity of itch (pruritus) due to AD was assessed using a horizontal NRS. Participants at specified time points were asked the following question: "How would you rate your itch due to AD at the worst moment during the previous 24 hours?" The scale ranged from 0-10, where 0= no itch and 10= worst itch imaginable. Higher scores indicated worse itch.
Percentage of Participants Achieving >=4 Points Reduction in Peak Pruritus Numerical Rating Scale (PP-NRS) From Baseline at Week 2, 4, 12, 16, 24, and 52 | Baseline, Week 2, 4, 12, 16, 24, and 52
  The severity of itch (pruritus) due to AD was assessed using a horizontal NRS. Participants at specified time points were asked the following question: "How would you rate your itch due to AD at the worst moment during the previous 24 hours?" The scale ranged from 0-10, where 0= no itch and 10= worst itch imaginable. Higher scores indicated worse itch.
Percentage of Participants Achieving 0 or 1 in Peak Pruritus Numerical Rating Scale (PP-NRS) From Baseline at Week 2, 4, 12, 16, 24, and 52 | Baseline, Week 2, 4, 12, 16, 24, and 52
  The severity of itch (pruritus) due to AD was assessed using a horizontal NRS. Participants at specified time points were asked the following question: "How would you rate your itch due to AD at the worst moment during the previous 24 hours?" The scale ranged from 0-10, where 0= no itch and 10= worst itch imaginable. Higher scores indicated worse itch.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (8):
- Taiwan (8):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital at Kaohsiung, Kaohsiung City
  - Taipei Medical University - Shuang Ho Hospital, New Taipei City
  - NTUH, Taipei
  - MacKay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Hospital Linkou, Taoyuan District

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7451114